CLINICAL TRIAL: NCT03855137
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Atogepant for the Prevention of Chronic Migraine (Progress)
Brief Title: Efficacy, Safety, and Tolerability of Atogepant for the Prevention of Chronic Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3101-303-002; 2018-004337-32 (EudraCT Number); NCT04961671 (obsolete NCT alias)
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Chronic Migraine
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received atogepant-matching placebo tablets, orally, twice daily (BID) for 12 weeks in a double-blind (DB) treatment period.
  Interventions: Drug: Placebo
- Atogepant 30 mg BID (Active Comparator): Participants received atogepant 30 mg tablet, orally, BID and atogepant-matching placebo tablets orally, BID for up to 12 weeks in a DB treatment period.
  Interventions: Drug: Atogepant 30 mg; Drug: Placebo
- Atogepant 60 mg QD (Active Comparator): Participants received atogepant 60 mg, orally, once daily (QD) along with atogepant-matching placebo 30 mg as morning dose followed by atogepant-matching placebo 30 mg and 60 mg as evening doses for up to 12 weeks in a DB treatment period.
  Interventions: Drug: Atogepant 60 mg; Drug: Placebo

INTERVENTIONS:
Drug: Atogepant 30 mg — Tablets containing 30 mg atogepant
  Arms: Atogepant 30 mg BID
Drug: Atogepant 60 mg — Tablets containing 60 mg atogepant
  Arms: Atogepant 60 mg QD
Drug: Placebo — 30 mg/60 mg tablets containing atogepant-matching placebo

SUMMARY:
This study evaluated the efficacy, safety and tolerability of atogepant in participants with chronic migraine. This study included a 12-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of chronic migraine (CM) consistent with a diagnosis according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3), 2018
* Age of the participant at the time of migraine onset < 50 years
* Confirmation of headache/migraine headache day frequency as follows:

  * History of, on average, ≥ 15 headache days per month in the 3 months prior to Visit 1 in the opinion of the investigator AND
  * >=15 headache days during the 4-week screening/baseline period per the electronic diary (eDiary) AND
  * >=8 days during the 4-week screening/baseline period that qualify as being a migraine day per the eDiary
* Participants must be using a medically acceptable and effective method of birth control during the course of the entire study

Exclusion Criteria:

* Has a history of migraine, accompanied by diplopia or decreased level of consciousness, or retinal migraine
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy
* History of an inadequate response to > 4 medications (2 of which have different mechanisms of action) prescribed for the prevention of migraine
* Woman is pregnant, planning to become pregnant during the course of the study, or currently lactating. Women of childbearing potential must have a negative urine pregnancy test at Visit 1 and Visit 2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (150):
- United States (41):
  - Barrow Neuro Institute /ID# 236776, Phoenix, Arizona
  - Baptist Health Center for Clinical Research /ID# 237361, Little Rock, Arkansas
  - California Headache and Balance Center /ID# 236246, Fresno, California
  - Wr-Pri Llc /Id# 236008, Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Newport Beach (Wake) /ID# 237692, Newport Beach, California
  - Schuster Medical Research Institute /ID# 236447, Sherman Oaks, California
  - Alpine Clinical Research Center /ID# 234346, Boulder, Colorado
  - George Washington University Medical Faculty Associates /ID# 238011, Washington D.C., District of Columbia
  - Accel Research Sites - St Petersburg Clinical Research Unit /ID# 237161, St. Petersburg, Florida
  - Accel Research Sites - Tampa Clinical Research Unit /ID# 237485, Tampa, Florida
  - Premiere Research Institute - Palm Beach /ID# 238192, West Palm Beach, Florida
  - NeuroTrials Research Inc. /ID# 237364, Atlanta, Georgia
  - Josephson-Wallack-Munshower Neurology - NE /ID# 238234, Indianapolis, Indiana
  - Collective Medical Research /ID# 236400, Prairie Village, Kansas
  - Ochsner Clinic Foundation /ID# 236543, Covington, Louisiana
  - Beth Israel Deaconess Medical Center /ID# 237540, Boston, Massachusetts
  - BTC of New Bedford /ID# 236384, New Bedford, Massachusetts
  - Clinical Research Institute, Inc /ID# 238299, Minneapolis, Minnesota
  - Headache Neurology Research Institute /ID# 236464, Ridgeland, Mississippi
  - Nevada Headache Institute /ID# 236420, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center /ID# 237444, Lebanon, New Hampshire
  - Albuquerque Clinical Trials, Inc /ID# 236853, Albuquerque, New Mexico
  - Albany Medical Center Rheumatology /ID# 236540, Albany, New York
  - Dent Neurosciences Research Center, Inc. /ID# 237040, Amherst, New York
  - Headache Wellness Center /ID# 236431, Greensboro, North Carolina
  - Raleigh Neurology Associates /ID# 237141, Raleigh, North Carolina
  - Stetson-University of Cincinnati /ID# 236453, Cincinnati, Ohio
  - Abington Neurological Associates - Abington /ID# 236258, Abington, Pennsylvania
  - Preferred Primary Care Physicians, Inc. /ID# 236439, Pittsburgh, Pennsylvania
  - WR-ClinSearch /ID# 238288, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 237478, Memphis, Tennessee
  - DiscoveResearch, Inc /ID# 236274, Bryan, Texas
  - Texas Neurology /ID# 236359, Dallas, Texas
  - University of Texas Southwestern Medical Center /ID# 236941, Dallas, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic /ID# 236395, Salt Lake City, Utah
  - J. Lewis Research, Inc. Foothill Family Clinic South /ID# 236297, Salt Lake City, Utah
  - Highland Clinical Research /ID# 237816, Salt Lake City, Utah
  - MedStar Georgetown Neurology /ID# 236324, McLean, Virginia
  - Sentara Neurology Specialists - Virginia Beach /ID# 234349, Virginia Beach, Virginia
  - Northwest Clinical Research Center /ID# 237581, Bellevue, Washington
  - Puget Sound Neurology /ID# 236321, Tacoma, Washington
- Australia (2):
  - Royal North Shore Hospital /ID# 237008, St Leonards, New South Wales
  - The Royal Melbourne Hospital /ID# 236859, Parkville, Victoria
- Canada (5):
  - CHAMP Clinic /ID# 236252, Calgary, Alberta
  - Vancouver Island Health Authority /ID# 238053, Victoria, British Columbia
  - Ottawa Headache Centre Research Inc /ID# 236432, Ottawa, Ontario
  - Clinique des cephalees de Montreal /ID# 236266, Montreal, Quebec
  - Montreal Neurological Institut /ID# 236329, Montreal, Quebec
- China (16):
  - Peking University Third Hospital /ID# 238150, Beijing, Beijing Municipality
  - Chinese PLA General Hospital /ID# 238237, Beijing, Beijing Municipality
  - Guangzhou First People's Hospital /ID# 236510, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University /ID# 238133, Guangzhou, Guangdong
  - Hubei General Hospital /ID# 236486, Wuhan, Hebei
  - The First Affiliated Hospital of Zhengzhou University /ID# 237025, Zhengzhou, Henan
  - Jiangsu Province Hospital /ID# 237846, Nanjing, Jiangsu
  - The Second Hospital of Jilin University /ID# 236520, Changchun, Jilin
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 237847, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University /ID# 236529, Taiyuan, Shanxi
  - The second Affiliated hospital of Zhejiang University school of Medicine /ID# 238260, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 236500, Hangzhou, Zhejiang
  - Beijing Friendship Hospital /ID# 237264, Beijing
  - The Second Hospital of Soochow University /ID# 234296, Suzhou
  - Tianjin Huanhu Hospital (THH) /ID# 236524, Tianjin
  - Tongji Hospital Tongji Medical College of HUST /ID# 237835, Wuhan
- Czechia (9):
  - NEUROHK s.r.o. /ID# 236290, Hradec Králové
  - BRAIN-SOULTHERAPY s.r.o. /ID# 236380, Kladno
  - CCR Ostrava, s.r.o. /ID# 234291, Ostrava
  - CLINTRIAL s.r.o. /ID# 237793, Prague
  - CCR Prague s.r.o. /ID# 236250, Prague
  - CCR Czech a.s /ID# 236249, Prague
  - Thomayerova nemocnice /ID# 237175, Prague
  - FORBELI s.r.o. /ID# 236427, Prague
  - NeuroMed Zlin s.r.o. /ID# 236416, Zlín
- Rigshospitalet Glostrup /ID# 236411, Glostrup Municipality, Capital Region, Denmark
- France (4):
  - AP-HM - Hopital de la Timone /ID# 236285, Marseille, Bouches-du-Rhone
  - CH Annecy Genevois Site Annecy /ID# 236385, Pringy, Haute-Savoie
  - Hôpital Pierre Wertheimer /ID# 236969, Bron
  - CHU Gabriel Montpied /ID# 237323, Clermont-Ferrand
- Germany (7):
  - Charite Universitaetsklinikum Berlin - Campus Virchow /ID# 237256, Berlin
  - Praxis Dr. Gendolla /ID# 236311, Essen
  - Universitaetsklinikum Essen /ID# 237209, Essen
  - CTC North GmbH & Co. KG /ID# 236328, Hamburg
  - Vitos Orthopaedische Klinik Kassel gemeinnuetzige GmbH /ID# 236723, Kassel
  - Schmerzklinik Kiel /ID# 236444, Kiel
  - LMU Klinikum Campus Grosshadern /ID# 236293, München
- Italy (6):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico /ID# 237492, Bari
  - Azienda Ospedaliero Universitaria Careggi /ID# 237598, Florence
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 237291, Milan
  - AOU Universita degli Studi della Campania Luigi Vanvitelli /ID# 236361, Napoli
  - Universita di Pavia /ID# 236363, Pavia
  - IRCCS San Raffaele Pisana /ID# 236552, Rome
- Japan (23):
  - Takanoko Hospital /ID# 234564, Matsuyama, Ehime
  - Fukuiken Saiseikai Hospital /ID# 236794, Fukui-shi, Fukui
  - Higashi Sapporo Neurology and Neurosurgery Clinic /ID# 234549, Sapporo, Hokkaido
  - Konan Medical Center /ID# 236230, Kobe, Hyōgo
  - Atsuchi Neurosurgical Hospital /ID# 234779, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 237595, Isehara-shi, Kanagawa
  - Fujitsu Clinic /ID# 237443, Kawasaki-shi, Kanagawa
  - Umenotsuji Clinic /ID# 234495, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 234496, Sendai, Miyagi
  - Saitama Medical University Hospital /ID# 237019, Iruma-gun, Saitama
  - Saitama Neuropsychiatric Institute /Id# 234550, Saitama-shi, Saitama
  - Japanese Red Cross Shizuoka Hospital /ID# 234372, Shizuoka, Shizuoka
  - Dokkyo Medical University Hospital /ID# 236810, Shimotsuga-gun, Tochigi
  - Niwa Family Clinic /ID# 234552, Chofu-shi, Tokyo
  - Tokyo Headache Clinic /ID# 234555, Shibuya-ku, Tokyo
  - Keio University Hospital /ID# 237210, Shinjuku-ku, Tokyo
  - Nagaseki Headache Clinic /ID# 234561, Kai-shi, Yamanashi
  - DOI Internal Medicine-Neurology Clinic /ID# 234562, Hiroshima
  - Hiroshima Neurology Clinic /ID# 234563, Hiroshima
  - Tanaka Neurosurgical clinic /ID# 234760, Kagoshima
  - Tatsuoka Neurology Clinic /ID# 234782, Kyoto
  - Tominaga Hospital /ID# 234781, Osaka
  - Shinagawa Strings Clinic /ID# 234780, Tokyo
- Poland (8):
  - Solumed Centrum Medyczne /ID# 236452, Poznan, Greater Poland Voivodeship
  - NZOZ Vitamed /ID# 237041, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 236348, Krakow, Lesser Poland Voivodeship
  - Centrum Leczenia Padaczki i Migreny /ID# 236386, Krakow, Lesser Poland Voivodeship
  - Indywidualna Praktyka Lekarska dr hab. med. Anna Szczepanska-Szerej /ID# 236289, Lublin, Lublin Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 237077, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp. z o.o. /ID# 237343, Katowice, Silesian Voivodeship
  - EuroMedis sp. z o.o. /ID# 236417, Szczecin, West Pomeranian Voivodeship
- Russia (5):
  - Kazan State Medical University /ID# 236298, Kazan', Tatarstan, Respublika
  - State Autonomous Healthcare Institution Republican Clinical Neurology Centre /ID# 236354, Kazan', Tatarstan, Respublika
  - University Headache Clinic /ID# 236371, Moscow
  - Clinics Chaika /ID# 236394, Moscow
  - Central Clinical Hospital RZHD Medicine /ID# 237024, Moscow
- South Korea (7):
  - Dongtan Sacred Heart Hospital /ID# 238097, Hwaseong, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 237754, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 237839, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital /ID# 237120, Busan
  - Nowon Eulji Medical Center, Eulji University /ID# 236306, Seoul
  - Seoul National University Hospital /ID# 237786, Seoul
  - Samsung Medical Center /ID# 237785, Seoul
- Spain (8):
  - Hospital Clínico Universitario de Santiago-CHUS /ID# 237623, Santiago de Compostela, A Coruna
  - CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 237645, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron /ID# 236467, Barcelona
  - Hospital Universitario Virgen del Rocio /ID# 237106, Seville
  - Hospital Clinico Universitario de Valencia /ID# 237400, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 237087, Valencia
  - Hospital Clinico Universitario de Valladolid /ID# 234406, Valladolid
  - Hospital Clinico Universitario Lozano Blesa /ID# 237373, Zaragoza
- Stortorgets Neurologmottagning /ID# 236454, Helsingborg, Sweden
- Taiwan (5):
  - Kuang-Tien General Hospital /ID# 236309, Taichung
  - Tainan Sin Lau Hospital /ID# 236358, Tainan
  - Chi-Mei Medical Center /ID# 236724, Tainan
  - Taipei Veterans General Hosp /ID# 237236, Taipei
  - Tri-Service General Hospital /ID# 237657, Taipei
- United Kingdom (2):
  - Walton Centre /ID# 236468, Liverpool
  - King's College Hospital NHS Foundation Trust /ID# 236301, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Schlachter L, Stodtmann S, Voelkner A, Jonsson F, Lagraauw HM, Boinpally RR. Population Pharmacokinetics of Atogepant for the Prevention of Migraine. Clin Pharmacokinet. 2025 Nov 12. doi: 10.1007/s40262-025-01566-5. Online ahead of print. PMID 41222899
- [Derived] UpToDate(R). Nurse Pract. 2023 Jul 1;48(7):16. doi: 10.1097/01.NPR.0000000000000072. No abstract available. PMID 40471213
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Lipton RB, Gandhi P, Tassorelli C, Reuter U, Harriott AM, Holle-Lee D, Gottschalk CH, Neel B, Liu Y, Guo H, Stokes J, Nagy K, Dabruzzo B, Smith JH. Early Improvements With Atogepant for the Preventive Treatment of Migraine: Results From 3 Randomized Phase 3 Trials. Neurology. 2025 Jan 28;104(2):e210212. doi: 10.1212/WNL.0000000000210212. Epub 2024 Dec 23. PMID 39715475
- [Derived] Peterlin BL, Bond DS, Ailani J, Dodick DW, Liu Y, De Abreu Ferreira R, Smith JH, Dabruzzo B, Goadsby PJ, Trugman JM. Weight loss with atogepant during the preventive treatment of migraine: A pooled analysis. Cephalalgia. 2024 Dec;44(12):3331024241299753. doi: 10.1177/03331024241299753. PMID 39648629
- [Derived] Gottschalk C, Gandhi P, Pozo-Rosich P, Christie S, Tassorelli C, Stokes J, Liu Y, Luo L, Nagy K, Trugman JM, Lipton RB. Effect of preventive treatment with atogepant on quality of life, daily functioning, and headache impact across the spectrum of migraine: Findings from three double-blind, randomized, phase 3 trials. Cephalalgia. 2024 Dec;44(12):3331024241300305. doi: 10.1177/03331024241300305. PMID 39648617
- [Derived] Goadsby PJ, Friedman DI, Holle-Lee D, Demarquay G, Ashina S, Sakai F, Neel B, Gandhi P, Dabruzzo B, Smith JH, Liu Y, Trugman JM. Efficacy of Atogepant in Chronic Migraine With and Without Acute Medication Overuse in the Randomized, Double-Blind, Phase 3 PROGRESS Trial. Neurology. 2024 Jul 23;103(2):e209584. doi: 10.1212/WNL.0000000000209584. Epub 2024 Jun 26. PMID 38924724
- [Derived] Pozo-Rosich P, Ailani J, Ashina M, Goadsby PJ, Lipton RB, Reuter U, Guo H, Schwefel B, Lu K, Boinpally R, Miceli R, De Abreu Ferreira R, McCusker E, Yu SY, Severt L, Finnegan M, Trugman JM. Atogepant for the preventive treatment of chronic migraine (PROGRESS): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Sep 2;402(10404):775-785. doi: 10.1016/S0140-6736(23)01049-8. Epub 2023 Jul 26. PMID 37516125
- [Derived] Boinpally R, McNamee B, Yao L, Butler M, McGeeney D, Borbridge L, Periclou A. A Single Supratherapeutic Dose of Atogepant Does Not Affect Cardiac Repolarization in Healthy Adults: Results From a Randomized, Single-Dose, Phase 1 Crossover Trial. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1099-1107. doi: 10.1002/cpdd.940. Epub 2021 May 4. PMID 33942560
- [Derived] Min KC, Kraft WK, Bondiskey P, Colon-Gonzalez F, Liu W, Xu J, Panebianco D, Mixson L, Dockendorf MF, Matthews CZ, Boinpally R. Atogepant Is Not Associated With Clinically Meaningful Alanine Aminotransferase Elevations in Healthy Adults. Clin Transl Sci. 2021 Mar;14(2):599-605. doi: 10.1111/cts.12917. Epub 2020 Nov 24. PMID 33142014
- See also: Related Information — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 778 participants were randomized in a 1:1:1 ratio to receive atogepant matching placebo, atogepant 30 mg twice daily (BID), or atogepant 60 mg once daily (QD) for up to 12 weeks in a double-blind (DB) treatment period followed by 4 week follow up (FU) period till end of study up to approximately 16 weeks.
Groups:
- Placebo: Participants received atogepant-matching placebo tablets, orally, BID for 12 weeks in a DB treatment period.
- Atogepant 60 mg QD: Participants received atogepant 60 mg, orally, QD along with atogepant-matching placebo 30 mg as morning dose followed by atogepant-matching placebo 30 mg and 60 mg as evening doses for up to 12 weeks in a DB treatment period.
Period: DB Treatment Period (Day 1 to Week 12)
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Started | 259 | 257 | 262
Safety Population (Safety population included all participants who received at least 1 dose of study intervention.) | 255 | 257 | 261
Modified Intent-to-Treat (mITT) Population (mITT population included all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, and 9 to 12) of eDiary data during the double-blind treatment period.) | 246 | 253 | 256
Off-treatment Hypothetical Estimand Population (Off-treatment hypothetical estimand population included all randomized participants who received ≥ 1 dose of study intervention, had an evaluable baseline period of eDiary data and had ≥ 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data during the study, regardless of whether on study treatment or off study treatment.) | 249 | 254 | 257
Completed | 230 | 231 | 233
Not Completed | 29 | 26 | 29
Not completed — Adverse Event | 10 | 13 | 9
Not completed — Lack of Efficacy | 5 | 2 | 1
Not completed — Withdrawal by Subject | 8 | 7 | 14
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Protocol Deviation | 5 | 3 | 2
Not completed — Non-compliance With Study Drug | 1 | 0 | 0
Period: FU Period (Week 12 to Week 16)
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Started (Out of 694 participants who completed the DB treatment period, only 517 participants continued the follow-up period.) | 169 | 179 | 169
Completed (Participants who completed the DB treatment period and rolled-over to other extension studies 3101-312-002 (NCT04686136), 3101-306-002 (NCT04437433),and 3101-311-002 (NCT04829747) were not required to enter the follow-up period.) | 161 | 170 | 165
Not Completed | 8 | 9 | 4
Not completed — Withdrawal by Subject | 5 | 6 | 3
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Protocol Deviation | 2 | 0 | 0
Not completed — Reason not Specified | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD | Total
Number analyzed (Participants) | 259 | 257 | 262 | 778
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (12.43) | 42.6 (11.89) | 41.7 (12.30) | 42.1 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 227 | 226 | 682
  Male | 30 | 30 | 36 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 6 | 31
  Not Hispanic or Latino | 246 | 245 | 256 | 747
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 95 | 95 | 93 | 283
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 7 | 8 | 9 | 24
  White | 154 | 151 | 157 | 462
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Monthly Migraine Days in mITT Population [Median (Full Range); unit: migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, and 9 to 12) of eDiary data during the double-blind treatment period.
  migraine days per month
    number analyzed (Participants) | 246 | 253 | 256 | 755
    (all) | 18.00 [8.0 to 28.0] | 18.00 [8.0 to 28.0] | 19.00 [9.0 to 28.0] | 18.2 [8.0 to 28.0]
Monthly Migraine Days in Off-Treatment Hypothetical Estimand Population [Median (Full Range); unit: migraine days per month] — A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days was defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Population: Off-treatment hypothetical estimand population included all randomized participants who received ≥ 1 dose of study intervention, had an evaluable baseline period of eDiary data and had ≥ 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data during the study, regardless of whether on study treatment or off study treatment.
  migraine days per month
    number analyzed (Participants) | 249 | 254 | 257 | 760
    (all) | 18.0 [8 to 28] | 18.0 [8 to 28] | 19.0 [9 to 28] | 18.3 [8 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days Across 12-Week Treatment Period in mITT Population
Description: Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days were defined as the total number of reported migraine days in diary divided by total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. Negative change from Baseline indicates improvement. A contrast from Mixed-effects model for repeated measures (MMRM) was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: Baseline to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, and 9 to 12) of eDiary data during the DB treatment period.
Measure: Median (Full Range); unit: migraine days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 246 | 253 | 256
migraine days per month | -4.63 [-21.9 to 9.7] | -7.13 [-27.0 to 7.7] | -7.27 [-22.3 to 12.9]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0001, Mixed Model Repeated Measures (MMRM) — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.41, 95% CI 2-sided [-3.48 to -1.33], Standard Error of Mean 0.547 — MMRM model=treatment group,visit,stratification by acute medication overuse,migraine prevention medication use and number of failures,region,and treatment group-by-visit as fixed factors and baseline and baseline-by-visit interaction as covariates
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -1.82, 95% CI 2-sided [-2.89 to -0.75], Standard Error of Mean 0.545 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days Across 12-Week Treatment Period in Off-Treatment Hypothetical Estimand Population
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Off-treatment hypothetical estimand population included all randomized participants who received ≥ 1 dose of study intervention, had an evaluable baseline period of eDiary data and had ≥ 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data during the study, regardless of whether on study treatment or off study treatment.
Measure: Median (Full Range); unit: migraine days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 249 | 254 | 257
migraine days per month | -4.65 [-21.9 to 9.7] | -7.00 [-27.0 to 7.7] | -7.19 [-22.3 to 12.9]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0001, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.24, 95% CI 2-sided [-3.31 to -1.16], Standard Error of Mean 0.547 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0024, MMRM; Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -1.66, 95% CI 2-sided [-2.72 to -0.59], Standard Error of Mean 0.544 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across 12-Week Treatment Period in mITT Population
Description: Participants recorded daily total duration of a headache in a diary. A headache day is any calendar day on which the participant experienced a headache pain lasting 2 hours or longer unless an acute headache medication was used after the start of the headache. The monthly (4-week) headache days were defined as the total number of reported headache days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of headache days during the last 28 days prior to the randomization date. Negative change from Baseline indicates improvement. A contrast from MMRM was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: headache days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 246 | 253 | 256
headache days per month | -4.26 [-23.7 to 6.7] | -7.16 [-26.3 to 9.0] | -6.71 [-22.3 to 9.0]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0001, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.32, 95% CI 2-sided [-3.38 to -1.26], Standard Error of Mean 0.541 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -1.87, 95% CI 2-sided [-2.93 to -0.81], Standard Error of Mean 0.538 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Mean Monthly Headache Days Across 12-Week Treatment Period in Off-Treatment Hypothetical Estimand Population
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: headache days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 249 | 254 | 257
headache days per month | -4.33 [-23.7 to 6.7] | -7.04 [-26.3 to 9.0] | -6.59 [-22.3 to 9.0]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0002, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.14, 95% CI 2-sided [-3.20 to -1.09], Standard Error of Mean 0.539 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0024, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -1.72, 95% CI 2-sided [-2.78 to -0.67], Standard Error of Mean 0.536 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across 12-Week Treatment Period in mITT Population
Description: An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) to treat an acute migraine. The monthly (4-week) acute medication use days were defined as the total number of reported acute medication use days in the diary divided by the total number of days with diary records during each 4-week period and multiplied by 28. Each 4-week period was averaged. Baseline is defined as the number of migraine days during the last 28 days prior to the randomization date. A negative change from Baseline indicates improvement. A contrast from MMRM was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 246 | 253 | 256
acute medication use days per month | -3.57 [-23.7 to 20.7] | -6.23 [-26.1 to 7.4] | -6.33 [-26.0 to 14.2]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0001, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.63, 95% CI 2-sided [-3.63 to -1.63], Standard Error of Mean 0.510 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.13, 95% CI 2-sided [-3.13 to -1.13], Standard Error of Mean 0.508 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Mean Monthly Acute Medication Use Days Across 12-Week Treatment Period in Off-treatment Hypothetical Estimand Population
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: acute medication use days per month
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 249 | 254 | 257
acute medication use days per month | -3.56 [-23.7 to 20.7] | -6.21 [-26.1 to 7.4] | -6.00 [-26.0 to 14.2]
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0002, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.52, 95% CI 2-sided [-3.52 to -1.53], Standard Error of Mean 0.507 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0024, MMRM; Least Squares Mean Difference = -2.09, 95% CI 2-sided [-3.09 to -1.10], Standard Error of Mean 0.505

7. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in 3-Month Average of Monthly Migraine Days in mITT Population
Description: Data is reported for 50% responders averaged at each 4-week period. 50% responders are participants with at least a 50 percent reduction from baseline in 3-month average of monthly migraine days. Participants recorded daily duration of migraine in a diary. A migraine day was any calendar day on which the participant experienced a migraine headache. The monthly (4-week) migraine days is equal to total number of reported migraine days in diary divided by total number of days with diary records in each 4-week period multiplied by 28. The values are rounded off to the first decimal value.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 246 | 253 | 256
percentage of participants | 26.0 | 42.7 | 41.0
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0003, Logistic regression — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.45 to 3.14] — Logistic regression for each atogepant group versus placebo with baseline monthly migraine days as covariate,stratification of region,acute medication overuse,migraine prevention medication and number of failures,treatment group as fixed factors
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, Logistic regression — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.38 to 3.00] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in 3-Month Average of Monthly Migraine Days in Off-Treatment Hypothetical Estimand Population
Description: as for outcome 7
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 249 | 254 | 257
percentage of participants | 26.5 | 42.1 | 40.1
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0006, Logistic regression — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.38 to 2.98] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, Logistic regression — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.29 to 2.79] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Migraine Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) Role Function-Restrictive Domain Score at Week 12 in Off-Treatment Hypothetical Estimand Population
Description: The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality of life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive (question numbers 1-7, score ranges 7 to 42) assesses how migraines limit one's daily social and work-related activities; Role Function Preventive (question numbers 8-11, score ranges 4 to 24) assesses how migraines prevent these activities; and the Emotional Function (question numbers 12-14, score ranges 3 to 18) domain assesses the emotions associated with migraines. Participants respond to items using a 6-point scale ranging from none of the time to all of the time. Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life. A contrast from MMRM was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: At Week 12
Population: Off-treatment hypothetical estimand population included all randomized participants who received ≥ 1 dose of study intervention, had an evaluable baseline period of eDiary data and had ≥ 1 evaluable postbaseline 4-week period (Weeks 1 to 4, 5 to 8, 9 to 12) of eDiary data during the study, regardless of whether on study treatment or off study treatment. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 225 | 229 | 236
score on a scale | 17.56 (21.901) | 25.73 (23.137) | 23.72 (24.335)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0006, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = 7.43, 95% CI 2-sided [3.77 to 11.09], Standard Error of Mean 1.864 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0024, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = 5.78, 95% CI 2-sided [2.15 to 9.41], Standard Error of Mean 1.848 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in Mean Monthly Performance of Daily Activities Domain Score of the AIM-D Across 12-Week Treatment Period in mITT Population
Description: The AIM-D is a 11-item patient-reported outcome (PRO) measure that assesses the impact of migraine on the performance of daily activities which include, 7 items: difficulty with household chores, errands, leisure activities at home, leisure or social activities outside the home, strenuous physical activities, concentrating, and thinking clearly and physical impairment; 4 items: difficulty walking, moving body, bending forward, moving head using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw performance of daily activities domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden). A contrast from MMRM was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: Baseline to Week 12
Population: mITT Population included all randomized participants who received at least 1 dose of study intervention, had an evaluable baseline period of eDiary data, and had at least 1 evaluable post-baseline 4-week period (Weeks 1 to 4, 5 to 8, and 9 to 12) of eDiary data during the DB treatment period. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 226 | 225 | 231
score on a scale | -9.80 (11.311) | -14.56 (13.042) | -13.90 (12.625)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0003, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -4.85, 95% CI 2-sided [-6.75 to -2.95], Standard Error of Mean 0.968 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0009, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -3.38, 95% CI 2-sided [-5.27 to -1.49], Standard Error of Mean 0.963 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Mean Monthly Physical Impairment Domain Score of the AIM-D Across 12-Week Treatment Period in mITT Population
Description: The AIM-D is a 11-item PRO measure that assesses the impact of migraine on the performance of daily activities which includes 7 items: difficulty with household chores, errands, leisure activities at home, leisure or social activities outside the home, strenuous physical activities, concentrating, and thinking clearly and physical impairment; 4 items: difficulty walking, moving body, bending forward, moving head using a 6-point rating scale where 0=not difficult at all, 1=a little difficult, 2=somewhat difficult, 3=very difficult, 4=extremely difficult, and 5=I could not do it at all. The raw physical impairment domain scores were transformed to 0-100 scale, with higher scores indicating greater impact of migraine (higher disease burden). A contrast from MMRM was used to obtain the average treatment effects across the 12-week treatment period.
Time Frame: Baseline to Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 226 | 225 | 231
score on a scale | -8.05 (10.923) | -12.34 (12.237) | -11.65 (12.172)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0003, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -4.19, 95% CI 2-sided [-5.95 to -2.43], Standard Error of Mean 0.897 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0025, MMRM — Adjusted p-value using graphical approach to control the overall type 1 error rate for multiple comparisons; Least Squares Mean Difference = -2.71, 95% CI 2-sided [-4.47 to -0.96], Standard Error of Mean 0.893 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in the Headache Impact Test (HIT-6) Total Score at Week 12 in Off-Treatment Hypothetical Estimand Population
Description: HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function. Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses - each of which is assigned a score ranging from 6 points (never) to 13 points (always). MMRM was used for the analyses.
Time Frame: At Week 12
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
Number analyzed (Participants) | 225 | 229 | 236
score on a scale | -5.18 (6.682) | -8.97 (8.475) | -7.97 (8.209)
Statistical Analysis 1: Comparison: Placebo vs Atogepant 30 mg BID; Test type: Superiority; p = 0.0006, MMRM; Least Squares Mean Difference = -3.30, 95% CI 2-sided [-4.67 to -1.93], Standard Error of Mean 0.697 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Atogepant 60 mg QD; Test type: Superiority; p = 0.0024, MMRM; Least Squares Mean Difference = -2.66, 95% CI 2-sided [-4.02 to -1.30], Standard Error of Mean 0.690 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (Up to approximately 16 weeks)
Description: All-Cause Mortality is reported for all randomized participants. Safety population included all participants who received at least 1 dose of study intervention and was used for serious adverse events and other adverse events.
Arm/Group | Placebo | Atogepant 30 mg BID | Atogepant 60 mg QD
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/257 | 0/262
Serious Adverse Events (participants affected / at risk) | 3/255 | 4/257 | 7/261
Other Adverse Events (participants affected / at risk) | 16/255 | 44/257 | 46/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | Atogepant 30 mg BID (N=257) | Atogepant 60 mg QD (N=261)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BENIGN OVARIAN TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=255) | Atogepant 30 mg BID (N=257) | Atogepant 60 mg QD (N=261)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 28 (28) | 26 (26)
NAUSEA (Gastrointestinal disorders) | 9 (9) | 20 (21) | 25 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT03855137/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03855137/SAP_001.pdf